CLINICAL TRIAL: NCT04255212
Title: Peripheral vs Central Pain Modulation Mechanisms Involved in Delayed Onset Muscles Soreness in Sport Climbers a Randomized Trial
Brief Title: Effects of Soft Tissue Treatment vs Mechanisms Explanation to Treat Delayed Onset Muscles Soreness Among Sport Climbers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giacomo Carta, Principal Investigator, Clinical Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 437038-15102019
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Central Nervous System Sensitization; Peripheral Nervous System Disorders; Muscle Soreness; Muscle Strength
Keywords: Sport climber; Delayed Onset Muscle Soreness; Central sensitization; Peripheral sensitization; Soft tissue treatment
MeSH Terms: conditions — Peripheral Nervous System Diseases; Myalgia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to their allocation that will not be communicated till the conclusion of the research. The outcome assessors are blinded to the allocation of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soft tissue treatment (Experimental): Participants will be treated with 5 minutes of deep tissue manual flossing on the proximal and medial aspect of the forearm of each side. Direction of the gentle repeated manual compressions and shifts will be proximal to distal or vicerversa depending on the symptom reduction reported by the participants. Subjects will be instructed to report immediately if the manual treatment starts to induce an increase in symptoms.
  Interventions: Other: Soft tissue treatment
- Mechaninsms explanation (Placebo Comparator): Participants will be instructed with a 10 minute lesson on mechanisms hypothesized to generate Delayed Onset Muscle Soreness. To trigger the most the bottom down pain modulation given by the placebo effect lesson will be concluded stressing the fact that DOMS have a good prognosis and that in a short amount of time they will be pain free and also that no drugs are effective to reduce pain intensity in DOMS condition suggesting them to stay physically active.
  Interventions: Other: Mechaninsms explanation
- Control group (Other): Participants will be asked to wait 10 minutes and to relax until the tests will be performed again.
  Interventions: Other: Control Group
- Neurodynamic treatment (Experimental): Participants will be asked to lay supine on a medical table and keep their arms relaxed. 30 repetitions of gentle upper limb nerves mobilization, performed through a combination of neck and arm physiological movements, will be administered with cycles of tensions and relaxation of 1/5 seconds for 3 minutes in total for each arm. Subjects will be instructed to report immediately if the manual treatment starts to induce an increase in symptoms
  Interventions: Other: Neurodynamic treatment

INTERVENTIONS:
Other: Soft tissue treatment — Participants will be asked to sit in front of a medical table with their forearms supinated and relaxed. 5 minutes of deep tissue manual flossing on the proximal and medial aspect of the forearm of each side will be administered by keeping the hands contact on the skin of the participants for all the treatment duration. Direction of the gentle repeated manual compressions and shifts will be proximal to distal or vicerversa depending on the symptom reduction reported by the participants. Stimuli frequencies will be about 0,2-03 Hz. Subjects will be instructed to report immediately if the manual treatment starts to induce an increase in symptoms
  Other Names: compression combined to longitudinal repeated mobilization of the forearm soft tissues
  Arms: Soft tissue treatment
Other: Mechaninsms explanation — Participants will be instructed with a 10 minutes lesson on mechanisms hypothesized to generate Delayed Onset Muscle Soreness. To trigger the most the bottom down pain modulation given by the placebo effect lesson will be concluded stressing the fact that DOMS have a good prognosis and that in a short amount of time they will be pain free and also that no drugs are effective to reduce pain intensity in DOMS condition suggesting them to stay physically active.
  Arms: Mechaninsms explanation
Other: Control Group — Participants will be asked to wait 10 minutes and to relax until the tests will be performed again.
  Arms: Control group
Other: Neurodynamic treatment — Participants will be asked to lay supine on a medical table and keep their arms relaxed. 30 repetitions of gentle upper limb nerves mobilization, performed through a combination of neck and arm physiological movements, will be administered with cycles of tensions and relaxation of 1/5 seconds for 3 minutes in total for each arm. Subjects will be instructed to report immediately if the manual treatment starts to induce an increase in symptoms
  Arms: Neurodynamic treatment

SUMMARY:
The aim of the present research is to define the effects of short manual treatment of soft tissues compared to mechanisms explaining in Delayed Onset Muscle Soreness (DOMS) among sport climbers and to address the mechanisms of peripheral and central sensitization involved in DOMS phenomena.

DETAILED DESCRIPTION:
Sport climbing is a growing success sport that will be debuting as an official discipline in the Tokyo 2020 Olympics game. They are used during competitions.

To practice this discipline, both dexterity in movement and extreme physical strength are needed to climb the sloping and vertical walls that are used during competitions.

The appearance of muscle pain induced by an unusual and strenuous physical activity (DOMS) is an extremely common factor in all sports activities that involves a maximum and repeated muscular effort. In the sport climbing practice this physiological phenomenon is common and occurs both in those who practice at as professional and amateur level. Numerous studies have shown that muscle pain is induced by physical activity and independent of damage to muscle fibers and classic inflammation of tissues. The phenomenon of DOMS is accompanied by hyperalgesia and allodynia during muscle contraction, these are conditions of irritation of the peripheral nervous system (SNP) and central nervous system (CNS), but today no evidence of such sensitization phenomena of the SNP and SNC has been provided. The presence of muscle pain is one of the main causes of impossibility to practice sports not only for those who practice sport climbing at a professional level, but for most amateur sportsmen. Thanks to the tools validated in the last decade, it is possible to study the involvement and awareness responses of the SNP and SNC with reliable and non-invasive techniques in the phenomenon of DOMS. Understanding the mechanisms underlying the appearance of the DOMS is today a primary priority for sports practice and for physical training for muscular effort both as a professional and amateur level.

Presence of peripheral and central sensitization in DOMS will be assessed and a three arm randomized controlled double blind multicentric study will be performed to assess the effects of treatment on peripheral tissues compared to pain mechanisms explanation. Healthy participants of both sexes will be assessed before DOMS, at 48 hours (the peak phase of symptoms) before and after treatment and at 96 hours when symptoms usually are in remission.

ELIGIBILITY:
Inclusion Criteria:

* Being explained all the associated risks and benefits of the research
* Sign the written informed consent

Exclusion Criteria:

* Significant neck or upper limbs pain (with Numeric Pain Rating Scale [NPRS] greater than 3/10)
* Pregnancy
* Recent neck or arm surgery or significant trauma in the preceding 3 months
* Cancer or inflammatory disorders,
* Spinal cord or cauda equina signs
* Widespread neurological disorders affecting the tone of upper limbs and neck muscles
* Underlying diseases, such as diabetes mellitus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Numeric Pain Rating Scale at one week | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  pain intensity will be tested asking the standardized question " on a scale from 0 to 10 when 0 is no pain and 10 is the worst pain ever rate the pain intensity you feel in this moment in the body part assessed"
Change from Baseline Mechanical allodynia at one week | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  The assessor thumb will be placed over the testing area and pressure will be applied for 10 s (Scholz et al., 2009). The pressure will be sufficient to indent the soft tissues and lead to skin blanching
Change from Baseline Wind-Up at one week | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  10 nociceptive standardized stimuli will be administered on the skin of the painful area involved by muscle soreness on the medial aspect of the proximal forearm
Change from Baseline Upper limb neurodynamic test at one week | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  The validated test to detect upper limb peripheral nervous system neuropathies involving physiological combined passive movements of the upper limb will be administered with the participant laying supine on a medical table.
Change from basaeline Muscle endurance (flexor digiturum profundis and superficialis) test at one week | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  subjects will be required to keep their body weight lifted from the ground, hanging as much time as possible with their fingers on a standardized metal bar

SECONDARY OUTCOMES:
Change from Baseline Forearm circumference | The test will be administered at baseline, before the first climbing training session, at 48 hours before and after treatment administration, and at 96 hours from baseline
  using a standardized measuring tape circumference of the forearm at a standardized distance from the medial epicondylus will be recorded
Change from post treatment Perceived Reported Outcome Measure at 48 hours follow-up as Likert scale | The test will be administered after treatment at 48 hours from baseline and at 96 hours from baseline
  A validated self administered 11 point Likert scale whit "0 Much Better and 10 Much Worse" will be fulfilled by participants to assess the degree of change in participant painful condition induced from the treatment administered.
Change from post treatment Perceived Reported Outcome Measure at 48 hours follow-up | The test will be administered after treatment at 48 hours from baseline and at 96 hours from baseline
  It will be administered a validated categorical self administered scale of perceived improvement that inquires the pain intensity perceived changes induced by the treatment received:
  "Since when did you start the treatment, can you describe your impression of how your painful condition has changed (limitation of physical activity, emotion and quality of life)?" No change, (or even worsened) Always the same, it is difficult to think of an improvement A little better, but not remarkable Sometimes better, but change isn't a real difference Moderately better, a slight and noticeable improvement Better, a decided improvement that constitutes a real difference A big and decisive improvement, and that makes the difference
Change from Baseline Body Chart at one week | The test will be administered before first training, at 48 hours before and after treatment administration, and at 96 hours from baseline
  Symptoms will be reported topographically using a validated pain drawing tool to collect information on the symptom area and on their intensity and behaviour
Change from Baseline Central Sensitization Inventory at 48 hours | The test will be administered at baseline and after 48 hours before treatment
  A validated self administered inventory on the central sensitizing phenomenon will be administered. It briefly consists in a 25 item questionnaire that inquires the presence of symptoms related to central sensitization
Perceived Health Status | The test will be administered at baseline
  Perceived Health status will be tested using a 11 point Likert scale from 0 equal to the worts and 100 equal to the best perceived health status and subjects will be asked to report with an x their actual condition.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, Msc, Principal Investigator — University of Turin, Italy
Locations (2):
- Italy (2):
  - Department of Biological and Clinical Science - University of Turin, Orbassano, TO
  - Centro Universitario Sportivo, Torino, TO

IPD SHARING:
Plan to Share IPD: Yes
We intend to share all data after publication of the research on a scientific journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediatelly after scientific paper publication all data will be shared
Access Criteria: Data will be avaliable Online at the URL reported above

REFERENCES:
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Chiarotto A, Viti C, Sulli A, Cutolo M, Testa M, Piscitelli D. Cross-cultural adaptation and validity of the Italian version of the Central Sensitization Inventory. Musculoskelet Sci Pract. 2018 Oct;37:20-28. doi: 10.1016/j.msksp.2018.06.005. Epub 2018 Jun 15. PMID 29966856
- [Background] Egloff N, Klingler N, von Kanel R, Camara RJ, Curatolo M, Wegmann B, Marti E, Ferrari ML. Algometry with a clothes peg compared to an electronic pressure algometer: a randomized cross-sectional study in pain patients. BMC Musculoskelet Disord. 2011 Jul 25;12:174. doi: 10.1186/1471-2474-12-174. PMID 21787399
- [Background] Jensen TS, Finnerup NB. Allodynia and hyperalgesia in neuropathic pain: clinical manifestations and mechanisms. Lancet Neurol. 2014 Sep;13(9):924-35. doi: 10.1016/S1474-4422(14)70102-4. PMID 25142459
- [Background] Mizumura K, Taguchi T. Delayed onset muscle soreness: Involvement of neurotrophic factors. J Physiol Sci. 2016 Jan;66(1):43-52. doi: 10.1007/s12576-015-0397-0. PMID 26467448
- [Background] Paulsen G, Mikkelsen UR, Raastad T, Peake JM. Leucocytes, cytokines and satellite cells: what role do they play in muscle damage and regeneration following eccentric exercise? Exerc Immunol Rev. 2012;18:42-97. PMID 22876722